CLINICAL TRIAL: NCT02660307
Title: A Randomized Controlled Trial With a Follow-up Evaluation of a Stress Reduction Program for Companies - PROGRESS
Brief Title: A Stress Reduction Program for Companies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de estudos em Atenção Plena (Other)
Collaborators: SESI (Serviço Social da Indústria) (Unknown)
Responsible Party: Principal Investigator, Stephen William Little Me, Principal Investigator, Centro de estudos em Atenção Plena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROGRESS
Record Dates: First submitted 2015-12-22; First posted 2016-01-21 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Stress
Keywords: stress; work; employees; mindfulness; depression; anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PROGRESS group (Experimental): this group received the intervention based in meditation in the first 8 weeks. They were instructed to practice at least 5 times a week for up to half an hour a day. During the second 8 week period this group were left to manage their practice on their own.
  Interventions: Other: PROGRESS group
- control group (Other): this group received no intervention in the first 8 weeks. During the second 8 week period, this group received the same intervention based in meditation that received PROGRESS group.
  Interventions: Other: PROGRESS group

INTERVENTIONS:
Other: PROGRESS group

SUMMARY:
This protocol proposes a well-being program based in stress reduction program for employees of a company.

objectives: To evaluate the effects of a stress reduction program with a specific orientation for workers and taught to them within their companies.

Methods: Participants with stress complaints were recruited and randomized into two groups: group 1 (G1) received the intervention while group 2 (G2) did not. Both groups were evaluated before the intervention (time 1 - T1); again after the eight weeks of the program for G1 (time 2 - T2); and then at the end of a second eight-week period during which G2 received the intervention and G1 was simply instructed to maintain the practice they had learned without further instruction (time 3- T3).

DETAILED DESCRIPTION:
Disorders resulting from chronic stress are some of the main causes of absenteeism and reduced productivity in companies. A number of successful stress management programs are based on the principle of mindfulness and may help individuals to relieve stress symptoms and to improve well-being and pro-social behavior. The objective of this study was to evaluate the feasibility and efficacy of a weekly one-hour stress reduction program adapted for companies and if the possible benefits would be sustained 8 weeks after the end of the program. Participants with stress complaints were recruited in two companies and they were randomized into two groups: in the first period of the study, group 1 (G1) N=23 received the intervention while group 2 (G2) N=18 did not. Both groups were evaluated before the intervention (time 1 - T1); again after the eight weeks of the program for G1 (time 2 - T2); and then at the end of a second eight-week period during which G2 received the intervention and G1 was simply instructed to maintain the practice they had learned without further instruction (time 3- T3).

ELIGIBILITY:
Inclusion Criteria:

* workers with stress complaints aging from 18 to 60 years. They also had to have at least 8 years of education.

Exclusion Criteria:

* participants with a history of psychiatric or neurological disorders or who were under psychological or psychiatric treatment during the period of the study, or with a history of substance abuse, with the exception of tobacco.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
changes in subjective symptoms of stress | baseline, 8 weeks and 16 weeks
  questionnaire for stress symptoms via 37 somatic symptoms and 19 psychological symptoms.

SECONDARY OUTCOMES:
changes in subjective depression symptoms | baseline, 8 weeks and 16 weeks
  questionnaire for depression symptoms, 21 items describing depression symptoms, each item in a scale from 0 to 3.
changes in anxiety symptoms | baseline, 8 weeks and 16 weeks
  questionnaire for anxiety symptoms, 21 items describing anxiety symptom, each item in a scale from 0 to 3.
changes in speed of perception and visual and motor response | baseline, 8 weeks and 16 weeks
  this test is the association of numbers and symbols lasting 2 minutes. This variable measure is a neuropsychological test and the data presentation are in total scores
changes in Mindful Awareness and attention | baseline, 8 weeks and 16 weeks
  in a scale from 1 to 6 the participant classifies how frequently or infrequently he/she becomes aware or mindful by contemplating the 15 described daily conditions provided
changes in psychiatric symptoms | baseline, 8 weeks and 16 weeks
  questionnaire for psychiatric symptoms with 20 questions about mental health

CONTACTS AND LOCATIONS:
Overall Officials: stephen Little Me, Principal Investigator — Centro de estudos em Atenção Plena

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lacerda SS, Little SW, Kozasa EH. A Stress Reduction Program Adapted for the Work Environment: A Randomized Controlled Trial With a Follow-Up. Front Psychol. 2018 May 9;9:668. doi: 10.3389/fpsyg.2018.00668. eCollection 2018. PMID 29867646